CLINICAL TRIAL: NCT01181934
Title: A Double-Blind, Placebo-Controlled, Randomized Three-Way Crossover Study to Investigate The Effect of Nicotine on Arousal, Standard Cognitive Tasks And Social Cognition in Young and Elderly Healthy Subjects
Brief Title: The Effect of Nicotine on Arousal, Cognition and Social Cognition in Young and Elderly Healthy Subjects.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Clinical Scientist/Director, Experimental Medicine, Janssen Pharmaceutica N.V., Belgium
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: CR017251
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia; Cognition Disorders
Keywords: symptomatic treatment; cognition; cognitive deficits; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- 001 (Experimental): A643 (nicotine) 1mg oromucosal nicotine spray- three times daily during each treatment period
  Interventions: Other: A643 (nicotine)
- 002 (Experimental): A643 (nicotine) 2mg oromucosal nicotine spray- three times daily during each treatment period
  Interventions: Other: A643 (nicotine)
- 003 (Placebo Comparator): placebo placebo - three times daily during each treatment period
  Interventions: Drug: placebo

INTERVENTIONS:
Other: A643 (nicotine) — 2mg oromucosal nicotine spray- three times daily during each treatment period
  Arms: 002
Drug: placebo — placebo - three times daily during each treatment period
  Arms: 003
Other: A643 (nicotine) — 1mg oromucosal nicotine spray- three times daily during each treatment period
  Arms: 001

SUMMARY:
This study in young and elderly healthy subjects will investigate the effect of nicotine on arousal, cognitive task and social cognition after acute dose administration.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor subject knows the name of the assigned drug), placebo-controlled, randomized (study drug assigned by chance), three-way-crossover trial (participants may receive different interventions sequentially during the trial) in young and elderly healthy volunteers. The three-way-crossover treatment phase will consist of three blinded treatment periods separated by a wash out period (the period allowed for the entire administered drug to be eliminated from the body) of 2 to 7 days. The study duration for each volunteer will be approximately 8 weeks. Each volunteer enrolled will be randomized to receive Treatment A (1mg nicotine per dosing), Treatment B (2mg nicotine per dosing) or Treatment C (placebo) during one of their treatment period. The study drug (nicotine or placebo) will be administered three times daily on Day 1 of each treatment phase as a mouth spray, separated 2 to 3 hours from each other (i.e. 0h; and 2 to 3h; and 4 to 6h post first dosing). Three different blocks of cognitive assessments will follow, one after each drug administration. Safety evaluations include adverse event monitoring, vital signs and clinical laboratory tests. Each volunteer participating will receive 3 identical study drug administrations per dosing day (2 to 3 hours from each other), resulting in an overall dose of 3 mg nicotine (Treatment A), 6 mg nicotine (Treatment B) or 0 mg nicotine (Treatment C) per dosing day. By the end of the study, after the 3-way crossover, each volunteer will have received 9 mg nicotine via mouth spray.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 and 30 years of age inclusive (Cohort 1 only)
* Man or woman between 60 and 75 years of age, inclusive (Cohort 2 only)
* Body mass index (BMI) between 18 and 35 kg/m2, inclusive (BMI = eight/height2)
* Women must be: postmenopausal (for at least 12 months), surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), abstinent (at the discretion of the investigator/per local regulations), or if sexually active, be practicing a highly effective method of birth control and must agree to continue to use the same method of contraception throughout the study
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at admission (each study period)
* Men must agree to use a condom at each sexual intercourse and to not donate sperm during the study and for 3 months after receiving the last dose of study drug. In addition, their female partners should also use an appropriate method of birth control for at least the same duration

Exclusion Criteria:

* Female volunteers who are pregnant or breastfeeding
* Clinically significant abnormal values for clinical chemistry, hematology or urinalysis at screening. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to the investigator, are acceptable. Values of alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 2 fold Upper Limit of Normal will be allowed
* Clinically significant abnormal physical examination, vital signs or 12-lead ECG at screening
* History of epilepsy or fits or unexplained black-outs
* Current dangerous or aggressive behavior
* Clinically significant history of drug and/or food allergies
* Recent history (within previous 6 months) of alcohol or drug abuse
* Significant history of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, bronchospastic respiratory disease, dyspnea, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, infection, or any other illness that the investigator considers clinically significant should exclude the subject (Subjects with well-controlled hypertension will be allowed to participate)
* Significant history of or current psychiatric or neurological illness
* Smoking cigarettes (or equivalent) or the use of nicotine based products, within 3 months prior to study drug administration. Current use of any medication for smoking cessation such as nicotine replacement therapy, bupropion or varenicline
* Positive urine screen for drugs of abuse at screening or admission

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-05; Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of nicotine on measures of arousal and event related potentials, especially the P50 auditory evoked potential, as well as standard cognitive tasks and social cognition. | 1 hour post dose

SECONDARY OUTCOMES:
Nicotine exposure | predose and 5 min post each dosing

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.